CLINICAL TRIAL: NCT03685708
Title: Response to the HEPLISAV-B Hepatitis B Vaccine in Treatment Naive Chronic Lymphocytic Leukemia (CLL) and CLL Treated With Bruton's -Tyrosine Kinase Inhibitor (BTK-I)
Brief Title: HEPLISAV-B Hepatitis B Vaccine in Chronic Lymphocytic Leukemia (CLL) and CLL Treated With Bruton's-Tyrosine Kinase Inhibitor (BTK-I)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 180145; 18-H-0145
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-06

CONDITIONS: Hepatitis; Safety and Tolerability
Keywords: Ibrutinib; Acalabrutinib; Immunology
MeSH Terms: conditions — Hepatitis | interventions — Heplisav-B

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Chronic Lymphocytic Leukemia Patients That Are Treatment Naïve (Experimental): Treatment naïve Chronic Lymphocytic Leukemia (CLL) or small lymphocytic lymphoma (SLL) patients will receive HEPLISAV-B (Hepatitis B Vaccine [Recombinant ], adjuvanted) vaccine - A series of 2 doses (0.5 ml each) will be given on a 0- and 3- month schedule via intramuscular injection.
  Interventions: Biological: HEPLISAV-B
- Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib (Experimental): Ibrutinib monotherapy for at least 6 months prior to administration of the first vaccine dose in patients with Chronic Lymphocytic Leukemia (CLL) or small lymphocytic lymphoma (SLL). Patients will receive HEPLISAV-B (Hepatitis B Vaccine [Recombinant ], adjuvanted) vaccine - A series of 2 doses (0.5 ml each) will be given on a 0- and 3- month schedule via intramuscular injection.
  Interventions: Biological: HEPLISAV-B
- Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib (Experimental): Acalabrutinib monotherapy for at least 6 months prior to administration of the first vaccine dose in patients with Chronic Lymphocytic Leukemia (CLL) or small lymphocytic lymphoma (SLL). Patients will receive HEPLISAV-B (Hepatitis B Vaccine [Recombinant ], adjuvanted) vaccine - A series of 2 doses (0.5 ml each) will be given on a 0- and 3- month schedule via intramuscular injection.
  Interventions: Biological: HEPLISAV-B

INTERVENTIONS:
Biological: HEPLISAV-B — HEPLISAV-B (Hepatitis B Vaccine [Recombinant ], adjuvanted) vaccine - A series of 2 doses (0.5 ml each) will be given on a 0- and 3- month schedule via intramuscular injection.

SUMMARY:
Background:

People with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) tend to get infections more easily. This is because their immune systems are weakened. Hepatitis B is a virus that can be transmitted when body fluids from an infected person enter the body of an uninfected person. This virus can be dangerous for people with leukemia and lymphoma. HEPLISAV-B is a new hepatitis B vaccine. Researchers want to see if it can protect people with CLL/SLL from getting hepatitis B.

Objective:

To learn how HEPLISAV-B works in people who have CLL or SLL.

Eligibility:

Adults 18 years and older with CLL (or SLL). They must be getting no treatment for their CLL, or getting ibrutinib or acalabrutinib for it.

Design:

This study lasts 6 months from the date of first vaccination.

Participants may be screened with:

Physical exam

Blood tests

Pregnancy test

Visit 1

Participants will get blood drawn and the study vaccine. It will be given as an injection. If they get any symptoms within 7 days of the vaccine, they will write them in a diary.

Visit 2

After 3 months, participants will come back to the NIH to get another blood draw and the second vaccine dose.

Visit 3

Participants will return 3 months after the second vaccine dose was given. They will have blood drawn.

DETAILED DESCRIPTION:
This study aims to determine the HEPLISAV-B hepatitis B vaccine efficacy in chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL) lymphocytic patients that are treatment naive or receiving Bruton s-tyrosine kinase inhibitor (BTK-I) therapy. (Note: Since CLL and SLL are considered the same disease, CLL/SLL will be referred to as CLL hereafter, unless otherwise specified).

Key Eligibility Criteria:

1. Diagnosis of CLL
2. Cohort 1: Treatment naive CLL or SLL patients
3. Cohort 2: Subjects must be receiving ibrutinib monotherapy for at least 6 months prior to administration of the first vaccine dose
4. Cohort 3: Subjects must be receiving acalabrutinib monotherapy for at least 6 months prior to administration of the first vaccine dose
5. No known active or past hepatitis B infection
6. No history of prior hepatitis B virus vaccination (approved or investigational)
7. Age greater greater than or equal to 18 years.
8. ECOG performance status of 0-1

Design:

Patients with CLL will enroll on the study for the purpose of determining the HEPLISAV-B vaccine efficacy in patients who are treatment naive ore receiving BTK-I therapy. A series of 2 doses of HEPLISAV-B will be given on a 0- and 3- month schedule by intramuscular injection. Subjects will be followed at regular intervals and receive serologic response assessment following completion of the HEPLISAV-B vaccine series (6 months after the first vaccine

administration).

Study Objectives:

Primary Objective:

a) Determine the rate of hepatitis B seroprotective titer achievement (anti-HBs greater than or equal to 10mIU/mL) following completion of the HEPLISAV-B 2-dose vaccine series (6 months after the first vaccine administration) in the following populations:

* CLL patients who are treatment naive (n=54)
* CLL patients receiving treatment with ibrutinib (n=27)
* CLL patients receiving treatment with acalabrutinib (n=27)

Secondary Objective:

a) Determine the safety and tolerability of the HEPLISAV-B vaccine among CLL patients who are treatment naive or receiving BTK-Is (ibrutinib or acalabrutinib).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of CLL/SLL which is made according to the updated criteria of the NCI Working Group.
* No known active or past hepatitis B infection
* No history of prior hepatitis B virus vaccination (approved or investigational)
* History of negative hepatitis B viral titers (negative HBsAg, HBsAb and HBcAb)
* Cohort 1: Treatment naive CLL patients
* Cohort 2: Subjects must be receiving ibrutinib monotherapy for at least 6 months prior to administration of the first vaccine dose
* Cohort 3: Subjects must be receiving acalabrutinib monotherapy for at least 6 months prior to administration of the first vaccine dose
* Age greater than or equal to 18 years.
* ECOG performance status of 0-1
* Able to comprehend the investigational nature of the protocol and provide informed consent.

EXCLUSION CRITERIA:

* Female patients who are currently pregnant.
* Any uncontrolled active systemic infection
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator s opinion, could compromise the subject s safety or put the study outcomes at undue risk
* History of severe allergic reaction to any component of HEPLISAV-B, including yeast
* Receive intravenous or subcutaneous immunoglobulin (IVIG) within 3 months prior to vaccination
* Concomitant use of immunosuppressive agents (e.g. steroids, radiotherapy, chemotherapy)
* Hereditary or acquired immunodeficiency syndrome unrelated to CLL
* Non-English speaking individuals will be excluded from the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher MT Pleyer, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Pleyer C, Ali MA, Cohen JI, Tian X, Soto S, Ahn IE, Gaglione EM, Nierman P, Marti GE, Hesdorffer C, Lotter J, Superata J, Wiestner A, Sun C. Effect of Bruton tyrosine kinase inhibitor on efficacy of adjuvanted recombinant hepatitis B and zoster vaccines. Blood. 2021 Jan 14;137(2):185-189. doi: 10.1182/blood.2020008758. PMID 33259596
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-H-0145.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 78 participants were assessed for eligibility and consented. 76 participants met eligibility criteria.
Period: Overall Study
Arm/Group | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib | Chronic Lymphocytic Leukemia Patients That Are Treatment Naïve
Started | 14 | 18 | 46
Completed | 13 | 16 | 37
Not Completed | 1 | 2 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Screen Fail | 0 | 1 | 1
Not completed — COVID 19 Pandemic | 1 | 1 | 6
Not completed — Disease Progression | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib | Chronic Lymphocytic Leukemia Patients That Are Treatment Naïve | Total
Number analyzed (Participants) | 14 | 18 | 46 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 22 | 37
  >=65 years | 5 | 12 | 24 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 20 | 29
  Male | 11 | 12 | 26 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 14 | 17 | 43 | 74
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 12 | 17 | 42 | 71
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HEPLISAV-B Seroprotective Titer (Anti-HBs 10mIU/mL)
Description: Determine the rate of hepatitis B seroprotective titer achievement (anti-HBs 10mIU/mL) following completion of the HEPLISAV-B 2-dose vaccine series (6 months after the first vaccine administration) among chronic lymphocytic leukemia (CLL) patients who are treatment naïve or receiving Bruton Tyrosine Kinase (BTK) inhibitors (Ibrutinib or Acalabrutinib).
Time Frame: 6 months after the first vaccine administration
Population: All participants that completed the 2 doses vaccine series and blood draws. 8 participants could not complete laboratory assessments due to COVID pandemic.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib | Chronic Lymphocytic Leukemia Patients That Are Treatment Naïve
Number analyzed (Participants) | 11 | 15 | 32
Participants | 0 | 1 | 9

2. Secondary Outcome: Number of Participants That Experienced Serious Adverse Events Following HEPLISAV-B Vaccine Among CLL Patients
Description: Determine the safety of the HEPLISAV-B vaccine among chronic lymphocytic leukemia (CLL) patients who are treatment naïve or receiving Bruton Tyrosine Kinase (BTK) inhibitors (Ibrutinib or Acalabrutinib).
Time Frame: 6 months after the first vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib | Chronic Lymphocytic Leukemia Patients That Are Treatment Naïve
Number analyzed (Participants) | 14 | 18 | 46
Participants | 0 | 0 | 1

3. Secondary Outcome: Number of Participants That Did Not Complete Study Due to Intolerance of the HEPLISAV-B Vaccine Among CLL Patients.
Description: Determine the tolerability of the HEPLISAV-B vaccine among chronic lymphocytic leukemia (CLL) patients who are treatment naïve or receiving Bruton Tyrosine Kinase (BTK) inhibitors (Ibrutinib or Acalabrutinib).
Time Frame: 6 months after the first vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib | Chronic Lymphocytic Leukemia Patients That Are Treatment Naïve
Number analyzed (Participants) | 14 | 18 | 46
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Events will be collected for 7 days following the first and second vaccine dose and followed until resolution
Description: All events whether volunteered by the subject, discovered by study personnel during questioning, or detected through physical examination, clinically significant laboratory test, or other means will be recorded.
Arm/Group | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib | Chronic Lymphocytic Leukemia Patients That Are Treatment Naïve
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/18 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/18 | 1/46
Other Adverse Events (participants affected / at risk) | 12/14 | 17/18 | 40/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib (N=14) | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib (N=18) | Chronic Lymphocytic Leukemia Patients That Are Treatment Naïve (N=46)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib (N=14) | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib (N=18) | Chronic Lymphocytic Leukemia Patients That Are Treatment Naïve (N=46)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1) | 9 (12)
Edema limbs (General disorders) | 3 (3) | 2 (4) | 10 (11)
Fatigue (General disorders) | 5 (11) | 8 (13) | 20 (36)
Flu like symptoms (General disorders) | 2 (4) | 0 (0) | 11 (19)
Injection site reaction (General disorders) | 2 (2) | 7 (9) | 8 (13)
Pain (General disorders) | 12 (32) | 16 (32) | 35 (98)
Bruising (Injury, poisoning and procedural complications) | 1 (3) | 3 (3) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vaccination site lymphadenopathy (General disorders) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (10) | 5 (9) | 19 (30)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 7 (8) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (6) | 8 (12) | 20 (26)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (7)
Fever (General disorders) | 0 (0) | 0 (0) | 4 (5)
Vaccination site lymphadenopathy (General disorders) | 0 (0) | 0 (0) | 4 (6)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 22 (35)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT03685708/Prot_SAP_000.pdf